CLINICAL TRIAL: NCT01359280
Title: Nurse Delivered Cell Phone Adherence Intervention
Brief Title: Nurse Delivered Cell Phone Adherence Intervention (Pick It UP)
Acronym: PIU
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Seth Kalichman, Professor, University of Connecticut
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: H10-332; 1R01NR012962-01 (NIH)
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Medication Adherence
Keywords: HIV; AIDS; Medication; Adherence
MeSH Terms: conditions — Medication Adherence; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Adherence Counseling + Text Messages (Experimental): Participants receive one office-based adherence counseling session and 4 phone-delivered counseling sessions focused on antiretroviral adherence strategies using a model of behavioral self regulation skills building. Participants also receive follow-up medication reminder text messages delivered by cell phone.
  Interventions: Behavioral: Adherence Counseling; Behavioral: Text Messages
- Adherence Counseling Only (Experimental): Participants receive one office-based adherence counseling session and 4 phone-delivered counseling sessions focused on antiretroviral adherence strategies using a model of behavioral self regulation skills building.
  Interventions: Behavioral: Adherence Counseling
- General Health Counseling Only (Placebo Comparator): Participants receive one office-based counseling session and 4 phone-delivered counseling sessions focused on general health and nutrition strategies using a model of behavioral self regulation skills building.
  Interventions: Behavioral: General Health Counseling
- General Health Messages + Text Messages (Placebo Comparator): Participants receive one office-based counseling session and 4 phone-delivered counseling sessions focused on general health and nutrition strategies using a model of behavioral self regulation skills building. Participants also receive follow-up medication reminder text messages delivered by cell phone.
  Interventions: Behavioral: General Health Counseling; Behavioral: Text Messages

INTERVENTIONS:
Behavioral: Adherence Counseling — 5 Sessions of theory-based medication adherence counseling
  Arms: Adherence Counseling + Text Messages; Adherence Counseling Only
Behavioral: General Health Counseling — 5 sessions of health improvement counseling
  Arms: General Health Counseling Only; General Health Messages + Text Messages
Behavioral: Text Messages — Daily medication regimen tailored adherence reminders delivered by cell phone
  Arms: Adherence Counseling + Text Messages; General Health Messages + Text Messages

SUMMARY:
Persistent adherence to antiretroviral therapy is necessary for the successful treatment of HIV infection. The proposed research will test a theory-based behavioral intervention that includes objectively monitoring HIV treatment adherence with corrective feedback delivered by cell phone. The study will also test the independent effects of an automated text message reminder system for sustaining adherence improvements. The intervention under study has utility for people living with HIV/AIDS In resource limited rural and urban settings.

DETAILED DESCRIPTION:
This study is testing a theory-based HIV treatment adherence intervention delivered by cell phone to patients in urban and rural areas. Adherence to antiretroviral (ART) medications is necessary to achieve HIV suppression and non-adherence can lead to treatment resistant genetic variants of HIV. People living with HIV/AIDS often experience difficulty sustaining high-levels of treatment adherence. Most factors that interfere with adherence are unanticipated and occur between clinical visits, including depression, side effects, substance use, and lapses in pharmacy refill. We will conduct a randomized clinical trial to test a cell phone-delivered theory-based medication adherence counseling intervention. The intervention is grounded in Self-Regulation Model and utilizes unannounced pill counts to monitor adherence and guide corrective feedback within the counseling context. Using pill count adherence information for counseling allows providers to detect and correct patient non-adherence within a time frame that can head off viral resistance. An experimental factorial design will test the effects of counseling and a text message reminder system as well the interaction of counseling and text message components with 600 men and women receiving HIV treatment. Following screening, informed consent and baseline assessments participants will be randomized to one of four intervention conditions:(a) self-regulation counseling + regimen tailored text message reminders; (b) self-regulation counseling only; (c) control counseling + regimen tailored text reminders; or (d) control counseling only. The study will therefore use a 2 (self-regulation counseling) x 2 (text message reminders) full factorial deign with participants followed for 9 months post-intervention. The primary endpoints are medication adherence assessed by unannounced pill counts and HIV RNA (viral load). This newly developed intervention strategy is grounded in Self-Regulation Theory and is designed for use in clinical settings with limited resources.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Currently taking HIV treatment medication with non-adherence

Exclusion Criteria:

* Under age 18
* Not HIV positive
* Not taking HIV treatment medications
* Adherent to HIV Medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Chart Abstracted Viral Load | 12 months retrospective
  Patient HIV viral load is abstracted from medical records at baseline and at 12-month retrospective follow-up.

SECONDARY OUTCOMES:
Unannounced Pill Count Adherence | Monthly
  Unannounced phone-based pill counts conducted monthly to obtain an objective measure of medication adherence

CONTACTS AND LOCATIONS:
Overall Officials: Seth C Kalichman, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States